CLINICAL TRIAL: NCT07352917
Title: A Prospective Phase II Open-Label Pilot Study Evaluating the Efficacy and Safety of Methotrexate in the Treatment of Severe Vulvar Lichen Sclerosus
Brief Title: Methotrexate for Severe Vulvar Lichen Sclerosus
Acronym: GRAVES-MTX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Dermatologica Arbache ltda (Other)
Responsible Party: Principal Investigator, SAMIR ARBACHE, Principal Investigator, Clinica Dermatologica Arbache ltda
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2025-12-19; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Vulvar lichen sclerosus; Quality of life; methotrexate
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-center, prospective, open-label, phase II pilot interventional trial with a single-group assignment. All enrolled participants will receive the same intervention, consisting of weekly subcutaneous methotrexate administration, and will be followed longitudinally for clinical and safety outcomes over a 12-month period. There will be no randomization, masking, or control group, consistent with the exploratory and feasibility-oriented nature of a pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Subcutaneous Methotrexate (Experimental): Participants allocated to this single study arm will receive subcutaneous injectable methotrexate, administered once weekly at a standardized initial dose of 12.5 mg. Dose adjustments may be made according to clinical response and safety monitoring, based on predefined protocol criteria. Folic acid supplementation will be administered on the day following the weekly methotrexate injection.
  Participants will be followed quarterly for a 12-month period. Subjective clinical efficacy outcomes will be assessed, along with objective analyses related to genital morphology, documented through standardized photographic records, as well as treatment safety outcomes, including clinical and laboratory assessments performed every three months.
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Methotrexate (MTX) — Subcutaneous injectable methotrexate administered once weekly, starting at a standardized initial dose of 12.5 mg per administration. Dose adjustments may be performed according to clinical response and safety monitoring, based on predefined protocol criteria. Folic acid supplementation will be administered on the day following the weekly methotrexate injection.

SUMMARY:
Vulvar lichen sclerosus is a chronic inflammatory skin disease affecting the vulva and genital region, which may cause intense pruritus, pain, burning sensations, and progressive scarring. In severe cases, the disease may lead to significant anatomical changes, sexual dysfunction, and a reduction in quality of life.

First-line treatment for vulvar lichen sclerosus consists of high-potency topical corticosteroids. Although many patients experience symptom relief, a considerable number of women continue to have persistent symptoms or progressive anatomical damage. For these patients, therapeutic options are limited.

MTX is an immunomodulatory medication that has been used for several decades in the treatment of inflammatory and autoimmune diseases. Previous clinical observations suggest that MTX may be beneficial for patients with severe or treatment-resistant vulvar lichen sclerosus; however, prospective clinical studies in this population remain scarce.

This prospective, open-label, phase II pilot study aims to evaluate the efficacy and safety of subcutaneous injectable MTX, administered once weekly at a standardized initial dose of 12.5 mg, in women with severe vulvar lichen sclerosus who have not responded adequately to standard topical therapy. Participants will receive treatment for 12 months, with regular clinical and laboratory monitoring.

The primary objective of the study is to assess whether treatment with MTX leads to improvement in symptoms and stabilization of vulvar skin changes, using patient-reported outcome measures and standardized clinical assessments. Secondary objectives include evaluation of treatment tolerability, adherence, and the occurrence of adverse events.

As a pilot study, this research is designed to generate preliminary data on feasibility, safety, and potential clinical benefit, which may guide future larger controlled studies and contribute to the development of evidence-based therapeutic strategies for women with severe vulvar lichen sclerosus.

DETAILED DESCRIPTION:
Vulvar lichen sclerosus is a chronic inflammatory dermatosis of the anogenital skin, characterized by epithelial thinning, dermal sclerosis, and progressive architectural distortion. In its severe form, the disease may present with persistent symptoms such as pruritus, pain, fissuring, and functional impairment, as well as irreversible vulvar anatomical changes.

Current standard management relies on the long-term use of high-potency topical corticosteroids. Although this approach is effective for many patients, a proportion of women with severe vulvar lichen sclerosus experience inadequate symptom control or continued progression of morphological changes.

For eligibility purposes, disease severity is defined according to the Vulvar Quality of Life Index (VQLI), a tool designed to measure the impact of vulvar disease on patients' quality of life. Clinical response over time will be assessed using the Clinical Scoring System for Vulvar Lichen Sclerosus. At present, evidence-based therapeutic guidance for severe vulvar lichen sclerosus remains limited.

Methotrexate (MTX) is an immunomodulatory agent with a long history of use in the treatment of inflammatory and autoimmune diseases. Its pharmacological properties, dosing strategies, and safety profile are well established in dermatology and rheumatology. Preliminary clinical observations suggest that MTX may offer benefit in selected patients with severe or treatment-refractory vulvar lichen sclerosus; however, prospective evaluations in this population remain scarce.

This study is designed as a prospective, open-label, phase II pilot clinical trial aimed at evaluating the feasibility, safety, and potential therapeutic effect of systemic MTX in women with severe vulvar lichen sclerosus refractory to standard topical therapy. The study adopts a single-arm design with longitudinal follow-up over a 12-month period.

Participants will receive subcutaneous injectable MTX administered once weekly, with a standardized initial dose of 12.5 mg. Dose adjustments may be performed based on clinical response and safety monitoring. Folic acid supplementation will be administered on the day following the weekly MTX injection to reduce the risk of adverse effects. Clinical and laboratory assessments will be performed every three months throughout the study period.

Treatment response will be assessed using the Clinical Scoring System for Vulvar Lichen Sclerosus. Subjective assessment will include quantification of symptom severity, specifically pruritus, burning sensation, and pain. Outcomes related to sexual discomfort will be recorded descriptively.

Objective assessment will be based on evaluation of vulvar morphological changes using structured criteria supported by standardized photographic documentation. A variable number of images will be obtained, with a minimum of two photographs per participant (baseline and month 12), and additional photographs may be obtained every three months during follow-up. All images will be reviewed by independent evaluators.

Safety outcomes will include systematic recording of adverse events, laboratory abnormalities, and treatment discontinuations throughout the study period.

The planned sample size of 12 participants was defined based on the exploratory and pilot nature of the study, with the primary objective of assessing feasibility, safety, and outcome variability rather than demonstrating definitive efficacy. Methodological guidance supports this sample size as sufficient to inform the design of future larger studies, particularly in the context of a low-prevalence condition and limited prior prospective data.

Methotrexate has been prescribed for several decades in the management of inflammatory and autoimmune diseases, with a well-characterized safety profile. Contemporary evidence suggests that certain historically perceived risks may be lower when modern dosing strategies and standardized monitoring protocols are applied. Consensus-based dermatologic guidelines support the safe use of low-dose weekly subcutaneous MTX when appropriate patient selection, folic acid supplementation, and rigorous clinical and laboratory monitoring are implemented. Known adverse effects, including hepatic, hematologic, and gastrointestinal toxicity, will be monitored according to established protocols.

As an exploratory pilot study, this trial is not designed to establish definitive efficacy. Its primary purpose is to assess protocol feasibility, characterize safety and tolerability, and generate preliminary clinical data to inform the design of future controlled studies and contribute to the development of evidence-based systemic treatment strategies for women with severe vulvar lichen sclerosus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of genital lichen sclerosus et atrophicus (vulvar, perineal, or perianal);
* Histopathological diagnosis of genital lichen sclerosus et atrophicus;
* Disease severity defined according with a score above 24 on the Vulvar Quality of Life Index (VQLI);
* Failure of symptom regression or progressive genital deformity after at least 3 months of treatment with a high-potency topical corticosteroid;
* Normal baseline laboratory evaluation, including complete blood count, liver and kidney function tests, and negative serologies for HIV and hepatitis B and C;
* For women of childbearing potential, a negative pregnancy test at screening.

Exclusion Criteria (assessed before signing the Informed Consent Form):

* Lack of full mental or psychiatric capacity;
* Need for assistance from a third party (legal guardian) to participate in the study;
* Significant difficulty in understanding or expressing oneself in Portuguese;
* Unavailability or inability to complete Likert-scale questionnaires;
* Inability to comply with study requirements, including adherence to the treatment schedule and attendance at follow-up visits;
* Unrealistic expectations regarding treatment benefits or the possibility of adverse effects;
* Intention to become pregnant during the study period;
* Refusal to adopt at least one adequate contraceptive method (hormonal or barrier) in women of childbearing potential;
* Poor adherence to the commitment to abstain from alcoholic beverages;
* Uncontrolled autoimmune comorbidities;
* Refusal to sign the Informed Consent Form after adequate explanation and clarification of doubts;
* Any indication of inability to comply with the conditions established in the research protocol. Decisions will be made to ensure participant safety and study integrity, with appropriate communication regarding the reasons for exclusion.

Exclusion Criteria (assessed after signing the Informed Consent Form):

* Elevation of liver enzymes above normal limits or impaired renal function during laboratory monitoring. Exclusion refers to discontinuation of the experimental intervention; however, the participant will continue to receive comprehensive medical follow-up as needed;
* Pregnancy. The participant will be withdrawn from the study intervention and referred for obstetric care, while continuing to receive medical follow-up;
* Lack of cooperation, failure to attend scheduled follow-up visits, or failure to undergo required laboratory monitoring;
* Any other condition that limits the participant's ability to comply with study procedures, as determined by the responsible investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in vulvar symptom severity | 12 months
  Change in vulvar symptom severity from baseline to 12 months, assessed using the total symptom score of the Clinical Scoring System for Vulvar Lichen Sclerosus (symptom domains only), as described by Günthert et al. (J Sex Med. 2012;9:2342-2350). The total score ranges from 0 to 30 points and is calculated by summing the items within the symptom domain, yielding a single aggregated value per assessment. Higher scores indicate greater symptom severity. Symptoms related to sexual discomfort or pain during sexual activity are not included in the primary outcome score and will be recorded separately and reported descriptively.

SECONDARY OUTCOMES:
Change in vulvar morphology | 12 months
  Change in vulvar morphology score from baseline to 12 months, assessed using the total morphology score of the Clinical Scoring System for Vulvar Lichen Sclerosus as described by Günthert et al. (J Sex Med. 2012;9:2342-2350). The morphology score is a single aggregated score, ranging from 0 to 12, with higher scores indicating greater morphological severity.
Change in vulvar-related quality of life | 12 months
  Change in vulvar-related quality of life from baseline to 12 months, assessed using the Vulvar Quality of Life Index (VQLI), as described by Saunderson et al. Australasian Journal of Dermatology 61.2 (2020): 152-157. Total VQLI scores range from 0 to 45, with higher scores indicating worse quality of life.
Safety and tolerability of methotrexate | 12 months
  Safety outcomes will include the incidence of adverse events, laboratory abnormalities, and treatment discontinuations throughout the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- DermoCentro, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding sharing of individual participant data (IPD) has not yet been made. This study is a pilot, single-center clinical trial with a small sample size involving sensitive clinical and photographic data. Any potential data sharing will be carefully considered after study completion, taking into account participant privacy, informed consent provisions, ethical approvals, and applicable data protection regulations. If data sharing is pursued, only de-identified data would be made available upon reasonable request and subject to appropriate approvals.

REFERENCES:
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharm Stat. 2005;4:287-291.
- [Background] Jasionowska S, Almadori A, Goble M, Langridge BJ, Iakovou D, Kamel F, McKenzie M, Mclean A, Boyle D, Zenner N, Swale V, Butler PEM. A systematic review of outcome measures evaluating treatment efficacy in vulval lichen sclerosus and evaluation of patients' priorities. Skin Health Dis. 2024 Jul 5;4(5):e422. doi: 10.1002/ski2.422. eCollection 2024 Oct. PMID 39355724
- [Background] Saunderson RB, Harris V, Yeh R, Mallitt KA, Fischer G. Vulvar quality of life index (VQLI) - A simple tool to measure quality of life in patients with vulvar disease. Australas J Dermatol. 2020 May;61(2):152-157. doi: 10.1111/ajd.13235. Epub 2020 Jan 27. PMID 31984477
- [Background] Gunthert AR, Duclos K, Jahns BG, Krause E, Amann E, Limacher A, Mueller MD, Juni P. Clinical scoring system for vulvar lichen sclerosus. J Sex Med. 2012 Sep;9(9):2342-50. doi: 10.1111/j.1743-6109.2012.02814.x. Epub 2012 Jul 3. PMID 22759453
- [Background] Ghafari-Saravi A, Foster E. Treatment of Refractory Vulvar Lichen Sclerosus With Methotrexate. J Low Genit Tract Dis. 2024 Apr 1;28(2):202-204. doi: 10.1097/LGT.0000000000000795. Epub 2024 Jan 10. PMID 38518219
- [Background] Cuellar-Barboza A, Bashyam AM, Ghamrawi RI, Aickara D, Feldman SR, Pichardo RO. Methotrexate for the treatment of recalcitrant genital and extragenital lichen sclerosus: A retrospective series. Dermatol Ther. 2020 Jul;33(4):e13473. doi: 10.1111/dth.13473. Epub 2020 Jun 23. No abstract available. PMID 32347617
- [Background] Urun M, Gursel Urun Y, Sarikaya Solak S. A case of extragenital linear lichen sclerosus along the lines of Blaschko responding to methotrexate. Acta Dermatovenerol Alp Pannonica Adriat. 2020 Sep;29(3):149-151. PMID 32975302
- [Background] Kreuter A, Tigges C, Gaifullina R, Kirschke J, Altmeyer P, Gambichler T. Pulsed high-dose corticosteroids combined with low-dose methotrexate treatment in patients with refractory generalized extragenital lichen sclerosus. Arch Dermatol. 2009 Nov;145(11):1303-8. doi: 10.1001/archdermatol.2009.235. PMID 19917961
- [Background] Nayeemuddin F, Yates VM. Lichen sclerosus et atrophicus responding to methotrexate. Clin Exp Dermatol. 2008 Aug;33(5):651-2. doi: 10.1111/j.1365-2230.2008.02721.x. Epub 2008 May 27. No abstract available. PMID 18507666
- [Background] Warren RB, Weatherhead SC, Smith CH, Exton LS, Mohd Mustapa MF, Kirby B, Yesudian PD. British Association of Dermatologists' guidelines for the safe and effective prescribing of methotrexate for skin disease 2016. Br J Dermatol. 2016 Jul;175(1):23-44. doi: 10.1111/bjd.14816. No abstract available. PMID 27484275
- [Background] Nguyen BT, Kraus CN. Vulvar Lichen Sclerosus: What's New? Cutis. 2024 Mar;113(3):104-106. doi: 10.12788/cutis.0967. No abstract available. PMID 38648581
- [Background] Hargis A, Ngo M, Kraus CN, Mauskar M. Systemic Therapy for Lichen Sclerosus: A Systematic Review. J Low Genit Tract Dis. 2024 Jan 1;28(1):84-90. doi: 10.1097/LGT.0000000000000775. Epub 2023 Nov 4. PMID 37924260
- [Background] Singh N, Mishra N, Ghatage P. Treatment Options in Vulvar Lichen Sclerosus: A Scoping Review. Cureus. 2021 Feb 24;13(2):e13527. doi: 10.7759/cureus.13527. PMID 33786234